CLINICAL TRIAL: NCT02760914
Title: Inflammatory Activity in Various Compartments of Adipose Tissue in Patients With Coronary Heart Disease
Brief Title: Adipose Tissue and Inflammation in Coronary Heart Disease
Acronym: ATICH
Status: Active, not recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Svein Solheim, MD, PhD, Oslo University Hospital
Other Study IDs: 2016/441
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Coronary Heart Disease
Keywords: adipose tissue; inflammatory mediators; gene expression
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — adipose tissue, whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Coronary heart disease: Patients with coronary heart disease undergoing planned coronary artery bypass surgery

SUMMARY:
The aims of the present project are to study possible differences in inflammatory gene expression and protein secretion in various compartments of adipose tissue being exposed during open cardiac surgery in patients with coronary heart disease undergoing coronary artery bypass surgery.

DETAILED DESCRIPTION:
The present study is observational with biochemical end-points to disclose inflammatory mechanisms in various compartments of adipose tissue in patients with coronary heart disease (CHD) compared to patients without significant CHD. Fifty patients with CHD undergoing coronary artery bypass surgery with open chest procedure will be included and 20 patients with valve disease without overt CHD undergoing open valve surgery will serve as a control group. No specific restrictions to inclusion other than lack of consent to participate after written and oral information are listed. In patients undergoing open heart surgery for CHD, representative peri-operative biopsies from epicardial, pericardial and subcutaneous fat will be gathered, carefully processed and deep-frozen to 80 degrees of frost for later analyses on histological/cellular components and on messenger ribonucleic acid for selected inflammatory variables. Simultaneously, blood samples (arterial blood at start of operation) will be collected, processed and deep-frozen at 80 degrees of frost for later analyses of relevant circulating inflammatory variables to correlation analyses with tissue samples, possibly also PaxGene tubes for messenger ribonucleic acid in circulating leukocytes.

The study will be conducted according to the Declaration of Helsinki, and in accordance with approval from the Regional Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary heart disease undergoing coronary artery bypass surgery

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with coronary heart disease undergoing planned coronary artery bypass surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Inflammasome-related proteins | At inclusion
  Inflammasome-related proteins (IL-18, IL-1b, NLRP3, Caspase, TLR4, IL-6, IL-6R, gp130), markers of remodeling (i.e. MMP-9, TIMP-1, PAI-1, Galectin, EMMPRIN), adipokines (i.e adiponectin, visfatin), other relevant pro-and anti-inflammatory cytokines (like TNF-alpha, IL-8, IL-12, IFN-gamma, MCP-1, IL-4, IL-10, TGF beta.) Relevant laboratory methods; qPCR (mRNA - all compartments + PAXGenetubes (leukocytes); Immunohistochemically; Circulating (where possible) (ELISAs and/or Multiplex). Results will be recorded in a database for further statistical analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Ingebjørg Seljeflot, Professor, Principal Investigator — Oslo University Hospital, Ullevål, Oslo, Norway
Locations (1):
- Svein Solheim, Oslo, Norway

REFERENCES:
- [Derived] Opstad TB, Papotti B, Akra S, Hansen CH, Braathen B, Tonnessen T, Solheim S, Seljeflot I. Sirtuin1, not NAMPT, possesses anti-inflammatory effects in epicardial, pericardial and subcutaneous adipose tissue in patients with CHD. J Transl Med. 2023 Sep 21;21(1):644. doi: 10.1186/s12967-023-04518-4. PMID 37730614